CLINICAL TRIAL: NCT00909883
Title: Foot Dystonia Treatment by Botulinum Toxin Injections in Parkinson Disease : Efficiency of Injections Made in Extrinsic Muscle (Flexor Digitorum Longus Muscle) Compared to Intrinsic Muscle (Flexor Digitorum Brevis or Quadratus Plantae Muscles)
Acronym: RBHP 2008
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Merz Pharmaceuticals (Industry)
Responsible Party: Pr Franck DURIF, CHU Clermont-Ferrand
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0051
Record Dates: First submitted 2009-05-19; First posted 2009-05-29 (Estimated); Last update posted 2011-03-25 (Estimated); Status verified 2011-03

CONDITIONS: Parkinson's Disease; Foot Dystonia
Keywords: Idiopathic Parkinson's disease; Foot (Tiptoe) dystonia; Botulinum Toxin; Muscles : Flexor digitorum longus/ Flexor digitorum brevis/ quadratus plantae
MeSH Terms: conditions — Parkinson Disease; Dystonia

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Botulinum Toxin: Xeomin — 45 patients with an Idiopathic Parkinson's disease and a foot dystonia. Double blind, randomized study
Drug: Placebo — Placebo injection

SUMMARY:
Foot dystonia is frequently observed in patients suffering from Parkinson'disease. It is characterized by an abnormal involuntary movement which is very uncomfortable (difficult to walk) and painful for the patient.

Botulinum toxin injections seem to be efficient to treat this dystonia. However studies on this topic are few and very imprecise (many muscle injected, especially the Flexor digitorum longus, different doses used, heterogeneous population with many types of dystonia included, open studies).

DETAILED DESCRIPTION:
Study progress :

After an inclusion visit, patients are randomized in one of the 3 following groups :

* First group (PL : placebo) :

  * J0 : Patient will receive 1 injection of placebo in the Flexor digitorum longus and 1 injection of placebo in the Flexor digitorum brevis or in the quadratus plantae
  * J+1month : First evaluation
  * J+3 months : Patient will receive again 1 injection of placebo in the Flexor digitorum longus and 1 injection of placebo in the Flexor digitorum brevis or in the quadratus plantae
  * J+4 months : Last evaluation
* Second group (ME : Extrinsic muscle)

  * J0 : Patient will receive 1 injection of Botulinum toxin (100U) in the Flexor digitorum longus and 1 injection of placebo in the Flexor digitorum brevis or in the quadratus plantae
  * J+1 month : First evaluation
  * J+3 months : Patient will receive again 1 injection of Botulinum toxin (100U) in the Flexor digitorum longus and 1 injection of placebo in the Flexor digitorum brevis or in the quadratus plantae
  * J+4 months : Last evaluation
* Third group (MI : Intrinsic muscle)

  * J0 : Patient will receive 1 injection of placebo in the Flexor digitorum longus and 1 injection of Botulinum toxin (100U) in the Flexor digitorum brevis or in the quadratus plantae
  * J+1 month : First evaluations
  * J+3 months : Patient will receive again 1 injection of placebo in the Flexor digitorum longus and 1 injection of Botulinum toxin (100U) in the Flexor digitorum brevis or in the quadratus plantae
  * J+4 months : Last evaluations

During injections (J0 and J+3M), we will measure the pain induced by injections (EVA) For each evaluation (J+1M and J+4M), following evaluations will be made: clinical improvement (CGI), dystonia evaluation (duration and severity, Burke scale), pain (EVA) and quality of life (PDQ39).

ELIGIBILITY:
Inclusion Criteria:

* Age : 30-75 years
* Patient with an idiopathic Parkinson's disease according to the criteria of the "Parkinson's Disease Society Brain Bank"
* Patient with unilateral tiptoe dystonia. Dystonia must be present more than 1h /day and induce difficulties to walk (severity index ≥ 3 (1 : light, 2 : moderate, 3 : severe, 4 : very severe)).
* Patients never treated with botulinum toxin or already treated for more than 6 months.
* Affiliation to social security
* Agreement of patients

Exclusion Criteria:

* Patients suffering of an atypical Parkinson syndrome
* Patient with a bilateral tiptoe dystonia
* Patients with contraindication to the botulinum toxin use
* Women without efficient contraception
* Person who participate to an other study

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
In a controlled double blind and randomized study, we want to show that intramuscular injections of botulinum toxin are beneficial to reduced dystonia and associated pain in patient with foot dystonia (compared to placebo injections). | one month after the injection of botulinum toxin/placebo

SECONDARY OUTCOMES:
Efficiency comparison of injections made in leg muscle (Flexor digitorum longus) between injections made directly in foot muscle (Flexor digitorum brevis or quadratus plantae) - Effects of injections on pain and quality of life. | one month after injections of placebo or Botulinum toxin

CONTACTS AND LOCATIONS:
Overall Officials: Franck Durif, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (4):
- France (4):
  - CHU Purpan, Toulouse, Toulouse
  - CHU Gabriel-Montpied, Clermont-Ferrand
  - Hôpital La Pitié Salpétrière, Paris
  - Hôpital Haut-Levêque, Pessac